CLINICAL TRIAL: NCT01010555
Title: In-vivo Wettability Grading and Assessment Study
Acronym: CIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P-368-C-104
Record Dates: First submitted 2009-11-09; First posted 2009-11-10 (Estimated); Results first posted 2011-05-30 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- lotrafilcon B (Active Comparator): Lotrafilcon B contact lens randomly assigned to one eye, with balafilcon A contact lens assigned to the fellow eye for contralateral wear. Both products to be worn on a daily wear basis for 4 weeks, after which participant will wear senofilcon A contact lens randomly assigned to one eye and enfilcon A contact lens in the fellow eye for an additional 4 weeks of daily wear.
  Interventions: Device: lotrafilcon B
- balafilcon A (Active Comparator): Balafilcon A contact lens randomly assigned to one eye, with lotrafilcon B contact lens assigned to the fellow eye for contralateral wear. Both products to be worn on a daily wear basis for 4 weeks, after which participant will wear senofilcon A contact lens randomly assigned to one eye and enfilcon A contact lens in the fellow eye for an additional 4 weeks of daily wear.
  Interventions: Device: balafilcon A
- senofilcon A (Active Comparator): Senofilcon A contact lens randomly assigned to one eye, with enfilcon A contact lens assigned to the fellow eye for contralateral wear. Both products to be worn on a daily wear basis for 4 weeks, after which participant will wear lotrafilcon B contact lens randomly assigned to one eye and balafilcon A contact lens in the fellow eye for an additional 4 weeks of daily wear.
  Interventions: Device: senofilcon A
- enfilcon A (Active Comparator): Enfilcon A contact lens randomly assigned to one eye, with senofilcon A contact lens assigned to the fellow eye for contralateral wear. Both products to be worn on a daily wear basis for 4 weeks, after which participant will wear lotrafilcon B contact lens randomly assigned to one eye and balafilcon A contact lens in the fellow eye for an additional 4 weeks of daily wear.
  Interventions: Device: enfilcon A

INTERVENTIONS:
Device: lotrafilcon B — Commercially marketed, silicone hydrogel, spherical contact lens
  Other Names: Air Optix
  Arms: lotrafilcon B
Device: balafilcon A — Commercially marketed, silicone hydrogel, spherical contact lens
  Other Names: PureVision
  Arms: balafilcon A
Device: senofilcon A — Commercially marketed, silicone hydrogel, spherical contact lens
  Other Names: Acuvue OASYS
  Arms: senofilcon A
Device: enfilcon A — Commercially marketed, silicone hydrogel, spherical contact lens
  Other Names: Avaira
  Arms: enfilcon A

SUMMARY:
The purpose of this study is to investigate the front surface wettability of soft contact lenses while on eye.

ELIGIBILITY:
Inclusion Criteria:

* is at least 17 years of age
* has read and signed an information consent letter
* is a current daily wear contact lens wearer
* has acceptable fit with the study lenses
* has had an ocular exam in the last two years
* other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* has any ocular disease
* has undergone corneal refractive surgery or is aphakic
* has any systemic disease affecting ocular health
* is pregnant or lactating
* other protocol-defined exclusion criteria may apply

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research: University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four participants were enrolled but not dispensed due to failing inclusion/exclusion criteria (2) and withdrawing consent (2). These participants are included in the Actual Enrollment and Baseline Characteristics calculations, but not Participant Flow.
Pre-assignment Details: This reporting group includes all enrolled and dispensed participants.
Groups:
- Lotrafilcon B/Balafilcon A, Then Senofilcon A/Enfilcon A: Lotrafilcon B contact lens randomly assigned to one eye, with balafilcon A contact lens assigned to the fellow eye for contralateral daily wear. Both products worn for 4 weeks, followed by senofilcon A contact lens randomly assigned to one eye, with enfilcon A contact lens assigned to the fellow eye for an additional 4 weeks of contralateral daily wear.
- Senofilcon A/Enfilcon A, Then Lotrafilcon b/Balafilcon A: Senofilcon A contact lens randomly assigned to one eye, with enfilcon A contact lens assigned to the fellow eye for contralateral daily wear. Both products worn for 4 weeks, followed by lotrafilcon B contact lens randomly assigned to one eye, with balafilcon A contact lens assigned to the fellow eye for an additional 4 weeks of contralateral daily wear.
Period: First Four Weeks of Wear
Arm/Group | Lotrafilcon B/Balafilcon A, Then Senofilcon A/Enfilcon A | Senofilcon A/Enfilcon A, Then Lotrafilcon b/Balafilcon A
Started | 11 | 10
Completed | 11 (One participant who completed Period 1 did not start Period 2. Relocation.) | 10 (One participant who completed Period 1 did not start Period 2. Non-compliance with visit schedule.)
Not Completed | 0 | 0
Period: Second Four Weeks of Wear
Arm/Group | Lotrafilcon B/Balafilcon A, Then Senofilcon A/Enfilcon A | Senofilcon A/Enfilcon A, Then Lotrafilcon b/Balafilcon A
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled subjects.
Arm/Group | Overall
Number analyzed (Participants) | 25
Age Continuous [Median (Full Range); unit: years] | 20.0 [18 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: On-eye Wettability
Description: On-eye wettability, as assessed at the 4-week visit by a masked observer from a video taken of the eye 5 minutes after lens insertion. On-eye wettability was recorded on a 5-point scale, with 0=excellent and 4=very poor.
Time Frame: 4 weeks of wear
Population: Analysis conducted per protocol, with exclusions due to reasons such as, major protocol deviations as determined by masked review; discontinuations; and/or missing responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lotrafilcon B; Balafilcon A; Senofilcon A; Enfilcon A: Commercially marketed, silicone hydrogel, spherical contact lens worn in one eye on a daily wear basis for 4 weeks.
Arm/Group | Lotrafilcon B | Balafilcon A | Senofilcon A | Enfilcon A
Number analyzed (Participants) | 19 | 19 | 19 | 19
units on a scale | 1.33 (1.01) | 2.11 (1.16) | 1.70 (1.09) | 2.07 (1.00)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for the duration of the trial: 166 days.
Description: This reporting group includes all enrolled and exposed participants.
Arm/Group | Lotrafilcon B | Balafilcon A | Senofilcon A | Enfilcon A
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No distribution of trial-specific information without express written permission of Director of Centre for Contact Lens Research.